CLINICAL TRIAL: NCT04716621
Title: Pain Management in Primary Care: A Randomized Controlled Trial of a Computerized Decision Support Tool
Brief Title: Computerized Decision Support Tool for Pain Management in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MJHS Institute for Innovation in Palliative Care (Other)
Collaborators: Pfizer (Industry); The Institute for Family Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 8408357
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early intervention (Experimental): Three sites received the Pain Management Support System for Primary Care (PMSS-PC) integrated into the Electronic Health Record.
  Interventions: Other: Early intervention
- Delayed intervention (Other): Delayed wait-list control group. Three additional sites received the intervention 6 months after the first arm.
  Interventions: Other: Delayed intervention

INTERVENTIONS:
Other: Early intervention — The Pain Management Support System for Primary Care (PMSS-PC) generated "best practice alerts" and gave clinicians access to a pain assessment template, measures of psychological distress and substance use, guidelines for drug and non-drug therapies, and facilitated referrals. At implementation, clinicians at the practices were offered in-person and virtual education through six webinars on best practices for pain.
  Arms: Early intervention
Other: Delayed intervention — Delayed wait-list control group. The second arm involved three additional sites receiving the PMSS-PC intervention 6 months after the first arm. Initial outcomes from the PMSS-PC Experimental Intervention arm were compared to those of this Wait-list Control arm.
  Arms: Delayed intervention

SUMMARY:
Chronic pain is highly prevalent, compromises quality of life, and increases care utilization. Primary care providers are challenged to provide effective treatments, use opioid therapy appropriately, and address the adverse consequences of pain. Technology-enabled decision support tools may provide a means to improve pain management in primary care.

The objective of this study was to evaluate a novel electronic health record (EHR)-based decision support tool-plus-education intervention for pain management in primary care.

DETAILED DESCRIPTION:
This randomized, wait-list controlled trial evaluated a novel EHR-based system for pain management among patients with chronic pain in six practices of a Federally Qualified Health Center network in New York.

ELIGIBILITY:
Inclusion Criteria:

1. Treated at the Institute for Family Health
2. Spoke English or Spanish
3. Received one or more prescriptions for an opioid or nonopioid analgesic during the past three months
4. Pain screening at the prior three office visits documented scores >3 on the 0-6 scale (FACES, Hicks et al., 2001).
5. Willingness to complete questionnaires three times
6. A commitment to return to the practice
7. Reachable by phone
8. No evidence of psychopathology or cognitive impairment severe enough to prevent informed consent or completing the survey instruments

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2013-11-11 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Worst Pain Intensity | From baseline to 6 months following intervention implementation
  Worst pain intensity score on the Brief Pain Inventory-Short Form. Scores range from 0-10, with higher scores indicating more severe worst pain intensity.
Average Pain Intensity | From baseline to 6 months following intervention implementation
  Average pain intensity score on the Brief Pain Inventory-Short Form. Scores range from 0-10, with higher scores indicating more severe average pain intensity.
Pain Interference with Function | From baseline to 6 months following intervention implementation
  Pain interference T-score, measured on the PROMIS Pain Interference Short Form. Higher scores indicate more pain interference with function.

SECONDARY OUTCOMES:
Worst Pain Intensity | From 6 to 12 months following intervention implementation
  Worst pain intensity score on the Brief Pain Inventory-Short Form. Scores range from 0-10, with higher scores indicating more severe worst pain intensity.
Average Pain Intensity | From 6 to 12 months following intervention implementation
  Average pain intensity score on the Brief Pain Inventory-Short Form. Scores range from 0-10, with higher scores indicating more severe average pain intensity.
Pain Interference with Function | From 6 to 12 months following intervention implementation
  Pain interference T-score, measured on the PROMIS Pain Interference Short Form. Higher scores indicate more pain interference with function.
Uptake of the PMSS-PC intervention tool | From baseline to 12 months following intervention implementation
  Use of the PMSS-PC decision support tool by primary care providers